CLINICAL TRIAL: NCT07392073
Title: Prospective Study of Changes in Peripheral Blood Effector Tumor Antigen-Specific T Cells for Predicting Efficacy of Chemoimmunotherapy in Non-Small Cell Lung Cancer
Brief Title: Peripheral Blood ETASTs for Predicting Efficacy of Chemoimmunotherapy in NSCLC
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Weibiao Zeng, Attending Physician, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: 20251026103020786-2
Record Dates: First submitted 2026-01-26; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Cancer; Lung Adenocarcinoma; Lung Squamous Cell Carcinoma; Stage IIIB Non-Small Cell Lung Cancer; Stage IV Non-Small Cell Lung Cancer; Advanced Non-Small Cell Lung Cancer
Keywords: Tumor Antigen-Specific T Cells; Effector T Cells; Circulating T Cells; Biomarkers; PD-1 Inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NSCLC Patients Receiving Chemoimmunotherapy: Patients with stage IIIB-IV non-small cell lung cancer receiving standard PD-1 inhibitor (such as pembrolizumab) combined with platinum-based chemotherapy (such as pemetrexed/carboplatin or paclitaxel/carboplatin regimen). Peripheral blood samples collected at baseline and after cycle 2 for ETAST quantification using CTT-NanoDT technology.
  Interventions: Diagnostic Test: Circulating Tumor-Specific T Cell Nanodetection Technology (CTT-NanoDT)

INTERVENTIONS:
Diagnostic Test: Circulating Tumor-Specific T Cell Nanodetection Technology (CTT-NanoDT) — Novel detection method for quantifying effector tumor antigen-specific T cells (ETASTs) in peripheral blood. PBMCs isolated from 5 mL peripheral blood are co-incubated with TATAN nanoparticles (whole tumor cell antigen-loaded nanoparticles, 50 μg/mL) for 48 hours. Activated ETASTs are identified and quantified by multi-color flow cytometry as CD3+CD8+IFN-γ+ and CD3+CD8+CD137+ double-positive cells. Quality control requires coefficient of variation (CV) < 5%.

SUMMARY:
The goal of this observational study is to explore whether changes in peripheral blood effector tumor antigen-specific T cells (ETASTs) can predict treatment outcomes in patients with advanced non-small cell lung cancer (NSCLC) receiving chemoimmunotherapy. The study aims to:

* Evaluate the relationship between ΔETAST levels (baseline to cycle 2) and progression-free survival
* Compare the predictive performance of ΔETASTs with traditional biomarkers (PD-L1, TMB)
* Assess whether ΔETASTs can identify patients more likely to benefit from PD-1 inhibitor plus chemotherapy

Participants will:

* Provide peripheral blood samples at baseline and after cycle 2 of treatment
* Undergo ETAST quantification using the CTT-NanoDT technology with TATAN nanoparticles
* Have standard tumor assessments every 2 cycles according to RECIST 1.1 criteria
* Be followed for progression-free survival and overall survival up to 24 months

DETAILED DESCRIPTION:
Non-small cell lung cancer (NSCLC) accounts for the majority of lung cancer cases globally. While immune checkpoint inhibitors (ICIs), particularly PD-1/PD-L1 inhibitors combined with platinum-based chemotherapy, have become standard first-line therapy for advanced NSCLC, only a subset of patients achieve clinical benefit. Current biomarkers including PD-L1 expression and tumor mutational burden (TMB) have limited predictive accuracy, creating an urgent need for more reliable biomarkers.

Tumor antigen-specific T cells (TASTs) are the actual effectors in ICI therapy, and successful ICI response depends on reactivation of these cells. However, detection of circulating tumor antigen-specific T cells (CTASTs) has been technically challenging due to their low frequency and heterogeneity in peripheral blood.

This study utilizes a novel Circulating Tumor-Specific T Cell Nanodetection Technology (CTT-NanoDT) developed by the research team. The technology employs Tumor Antigen-specific T cell Activating Nanoparticles (TATAN) loaded with whole tumor cell components to specifically activate and quantify effector TASTs (ETASTs) in peripheral blood.

Study Design:

This is a prospective, single-center, observational cohort study enrolling 80 patients with stage IIIB-IV NSCLC receiving standard PD-1 inhibitor plus platinum-based chemotherapy. Peripheral blood samples (5 mL) will be collected at two time points: baseline (T0, within 1 day before treatment initiation) and after completion of cycle 2 (T1, day 21 of cycle 2).

ETAST Detection Protocol:

1. PBMC isolation from peripheral blood using Ficoll density gradient centrifugation
2. Co-incubation of PBMCs with TATAN nanoparticles (50 μg/mL) for 48 hours at 37°C
3. Flow cytometric quantification of activated ETASTs defined as CD3+CD8+IFN-γ+ and CD3+CD8+CD137+ double-positive cells
4. Calculation of ΔETAST: [(ETASTs-T1 - ETASTs-T0) / ETASTs-T0] × 100%

Primary Endpoint:

Progression-free survival (PFS), defined as time from treatment initiation to first documented disease progression per RECIST 1.1 or death from any cause, assessed by independent radiology committee.

Secondary Endpoints:

1. Comparison of predictive performance (ROC curve AUC) between ΔETASTs and traditional biomarkers (PD-L1 TPS, TMB) using DeLong test
2. Objective response rate (ORR), overall survival (OS), disease control rate (DCR)
3. Treatment-related adverse events graded per CTCAE 5.0

Statistical Analysis:

Cox proportional hazards regression will assess the association between ΔETASTs and PFS. Patients will be stratified by median ΔETAST value into high and low change groups for survival comparisons using Kaplan-Meier curves and log-rank tests. Sample size of 80 provides 80% power to detect HR=0.42 with α=0.05, accounting for 15% dropout rate.

The study aims to establish ΔETASTs as a superior biomarker for predicting chemoimmunotherapy efficacy in NSCLC, potentially enabling precision patient selection and improving treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed stage IIIB-IV non-small cell lung cancer (NSCLC)
* Planned to receive PD-1 inhibitor combined with platinum-based chemotherapy (e.g., pembrolizumab + pemetrexed/carboplatin)
* Age 18-80 years
* ECOG performance status 0-1
* Expected survival ≥12 weeks
* Adequate bone marrow function: ANC ≥1.5×10⁹/L, PLT ≥100×10⁹/L
* Adequate hepatorenal function: Cr ≤1.5×ULN, ALT/AST ≤2.5×ULN
* At least one measurable lesion per RECIST 1.1 criteria
* Able to provide informed consent and comply with study procedures including serial blood sampling and imaging follow-up

Exclusion Criteria:

* No measurable disease per RECIST 1.1 criteria
* Tumor emergencies requiring immediate intervention (spinal cord compression, superior vena cava syndrome)
* Active untreated central nervous system metastases or leptomeningeal disease
* Prior treatment with immune checkpoint inhibitors within 4 weeks before enrollment
* Chronic use of immunosuppressive agents (e.g., corticosteroids >10 mg/day prednisone equivalent)
* Coagulation disorders (INR >1.5 or APTT >1.5×ULN) or ongoing anticoagulation therapy
* Poor vascular access precluding serial venipuncture (>5 mL per draw)
* Active hepatitis B (HBV DNA >2000 IU/mL), hepatitis C, or HIV infection
* Uncontrolled bacterial or fungal infection requiring systemic treatment
* Pregnancy or lactation
* Severe psychiatric disorder or communication barriers affecting informed consent or follow-up compliance

Withdrawal Criteria:

* Participant voluntary withdrawal with signed withdrawal statement
* Major protocol violations: failure to receive ≥2 cycles of planned chemoimmunotherapy; missing ≥2 critical timepoint blood samples (baseline, cycle 2)
* Uncontrollable grade ≥3 immune-related adverse events requiring permanent discontinuation of PD-1 inhibitor

Study Termination Criteria:

* Disease progression confirmed by imaging per RECIST 1.1 or clinical progression requiring radiotherapy
* Death or loss to follow-up >6 months
* Unacceptable grade 4 treatment-related toxicity
* Investigator determination that continued participation poses health risk to patient
* Study terminated by ethics committee for scientific or administrative reasons

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18-80 years with histologically confirmed stage IIIB-IV non-small cell lung cancer (adenocarcinoma or squamous cell carcinoma) with adequate performance status (ECOG 0-1) and organ function, receiving standard PD-1 inhibitor plus platinum-based chemotherapy as first-line or subsequent-line systemic treatment.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From treatment initiation to first documented disease progression or death, assessed up to 24 months
  Time from first dose of chemoimmunotherapy to first documented disease progression per RECIST 1.1 criteria (assessed by independent radiology committee) or death from any cause, whichever occurs first. Tumor assessments performed every 2 treatment cycles (approximately every 6 weeks).

SECONDARY OUTCOMES:
Change in Effector Tumor Antigen-Specific T Cells (ΔETASTs) | From baseline to after completion of cycle 2 (approximately day 42)
Predictive Performance Comparison: ΔETASTs vs. Traditional Biomarkers | At 6 months and 12 months after treatment initiation
Objective Response Rate (ORR) | Best overall response from treatment initiation through study completion, up to 24 months
  Proportion of patients achieving complete response (CR) or partial response (PR) per RECIST 1.1 criteria, assessed by independent radiology committee. Comparison between high vs. low ΔETAST groups.
Overall Survival (OS) | From treatment initiation to death from any cause, assessed up to 24 months
  Time from first dose of chemoimmunotherapy to death from any cause. Patients alive at end of study will be censored at last known alive date.
Incidence of Treatment-Related Adverse Events | From treatment initiation through 30 days after last treatment dose, up to approximately 24 months
  Incidence, type, and severity of adverse events related to chemoimmunotherapy, graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Particular focus on immune-related adverse events (irAEs) including pneumonitis, hepatitis, colitis, myocarditis, and endocrinopathies. Safety of blood sampling procedures also monitored.